CLINICAL TRIAL: NCT00607282
Title: Efficacy of Udenafil in Treatment of Erectile Dysfunction After Radical Resection for Sigmoid Colon and Rectal Cancer : a Randomized Controlled Trial
Brief Title: Efficacy of Udenafil After Radical Resection for Sigmoid Colon and Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-0610-038-004; SNUBH-GS-CR2
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Erectile Dysfunction; Sigmoid Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Erectile Dysfunction; Sigmoid Neoplasms; Rectal Neoplasms | interventions — udenafil; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): normal control group
  Interventions: Drug: Udenafil
- Udenafil (Experimental): oral administration of placebo for Udenafil (Dong-A Pharmaceutical co., Ltd, Seoul, Korea)
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Udenafil — oral administration of Udenafil, prn(2hours before anticipated intercourse, 8 times/months)
  Other Names: Zydena®, Dong-A Pharmaceutical co., Ltd, Seoul, Korea

SUMMARY:
The purpose of this study is to evaluate the efficacy of Udenafil (Zydena®, Dong-A Pharmaceutical co., Ltd, Seoul, Korea) in treatment of erectile dysfunction after radical resection for sigmoid colon and rectal cancer. In this study, the efficacy of Udenafil will be evaluated in treatment for patient with chronic erectile dysfunction, which developed after radical resection for sigmoid and rectal cancer and continues 12 months after the surgery.

DETAILED DESCRIPTION:
Post-pelvic surgery erectile dysfunction is of much interest to those performing sigmoid colon and rectal cancer surgery and their patients. Erectile dysfunction has been recognized to develop from damage to pelvic parasympathetic nerve, which are especially vulnerable during anterior rectal dissection. There may be also a contribution of psychological factors from the presence of stoma and fear of recurrent cancer. Recently, several studies reported that erectile dysfunction after rectal excision for rectal cancer was completely reversed or satisfactorily improved using oral erectile dysfunction drugs. Udenafil is a new phosphodiesterase type 5 (PDE 5) inhibitor for erectile dysfunction. Prior studies have also demonstrated a selectivity profile for udenafil that is similar to Sildenafil (viagra®) and tadalafil (Cialis®). But unlike tadalafil (Cialis®), it does not significantly inhibit the PDE11 isozyme and not produce significant myalgia. back pain, or leg pain.

This prospective, randomized study was designed to evaluate the efficacy of Udenafil treatment in treatment of erectile dysfunction after radical resection for sigmoid colon and rectal cancer. In order to conduct this study, enrolled patients will be randomly attributed to Udenafil group or placebo group.

ELIGIBILITY:
Inclusion Criteria:

* • Male patients between 19-70 years old in good general health

  * Patient willing to treat postoperative erectile dysfunction and participate in the study
  * Patient who understands and accepts to sign the informed consent form
  * Patient who received radical resection for sigmoid colon and rectal cancer. : erectile dysfunction was developed following operation, not preoperatively
  * Scores of IIEF-5 measured at 12 months after surgery is 16 or less

Exclusion Criteria:

* • Documented problem of preoperative erectile dysfunction

  * Past history of myocardial infarction, cerebrovascular disease
  * Under administration of nitrate
  * Liver dysfunction (SGOT or SGPT 100 IU/L or more)
  * Kidney dysfunction (serum Creatinine 3mg/dl or more)

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Improvement of erectile function using IIEF-5 (International Index of Erectile Function-5), SEP Q2, Q3 (Sexual Encounter Profile Q2,Q3), and GEQ (Global efficacy Question) | at 4 weeks after enrollment

SECONDARY OUTCOMES:
Improvement of erectile function using IIEF-5, SEP Q2,Q3, and GEQ | at 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, M.D., Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Surgery, Seoul National University Bundang Hospital, Seongnam, South Korea